CLINICAL TRIAL: NCT02373124
Title: Glutamatergic Modulation of Motivation Enhancement: A Pilot Feasibility Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Elias Dakwar, Assistant Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7051
Record Dates: First submitted 2015-01-30; First posted 2015-02-26 (Estimated); Results first posted 2019-04-24 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Cocaine Use Disorders
MeSH Terms: interventions — GluN2C-2D antagonist UBP145

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- open-label (Experimental): 52 minute infusion of NMDA antagonist
  Interventions: Drug: infusion of NMDA antagonist

INTERVENTIONS:
Drug: infusion of NMDA antagonist — 52 minute infusion
  Other Names: NMDA antagonist

SUMMARY:
This study evaluates the feasibility of a treatment paradigm that involves naturalistic cocaine use opportunities in the context of psychotherapy aimed at utilizing these opportunities therapeutically.

ELIGIBILITY:
Inclusion Criterion Method of Ascertainment

1. Active cocaine dependence with at least 8 days of use or at least 4 binges of large amounts (>$200/occasion) over the past 30 days, and displaying at least one positive utox during screening SCID, Psychiatric Interview, self-report, utox
2. Physically healthy Laboratory tests (urinalysis, blood chemistry, 12-lead ECG in normal limits), physical examination, self-reported medical history
3. No adverse reactions to study medications Subjects will be asked about previous exposure to ketamine and midazolam
4. 21-55 years of age Self-reported age, verification with legal identification
5. Capacity to consent and comply with study procedures, including sufficient proficiency in English A short written test about study procedures, SCID, psychiatric interview
6. Seeking treatment Psychiatric Interview, self-report

Exclusion Criterion Method of Ascertainment

1. Meets DSM IV criteria for current major depression, bipolar disorder, schizophrenia, any psychotic illness, including substance induced psychosis, and current substance-induced mood disorder with HAMD score > 12. Psychiatric Interview, SCID, HAMD
2. Physiological dependence on another substance, such as alcohol, opioids, or benzodiazepines, excluding caffeine, nicotine, and cannabis SCID, Psychiatric Interview
3. Delirium, Dementia, Amnesia, Cognitive Disorders, or Dissociative disorders SCID, Psychiatric Interview
4. Current suicide risk or a history of suicide attempt within the past year SCID, Psychiatric Interview
5. Pregnant or interested in becoming pregnant during the study period Blood and urine pregnancy testing, self-report
6. Any of the following cardiac conditions: clinically significant left ventricular hypertrophy, angina, clinically significant arrhythmia, or mitral valve prolapse Laboratory tests (12-lead ECG in normal limits), physical examination, self-reported medical history
7. Unstable physical disorders which might make participation hazardous such as end-stage AIDS, hypertension (>140/90), WBC < 3.5, active hepatitis or other liver disease with elevated transaminase levels (< 2-3 X upper limit of normal will be considered acceptable if PT/PTT is normal), renal failure (creat > 2, BUN >40), or untreated diabetes Physiological tests (urinalysis, blood chemistry, 12-lead ECG), physical examination, self-reported medical history
8. Previous history of ketamine or midazolam misuse or abuse, and a history of an adverse reaction/experience with prior exposure to cocaine, ketamine or midazolam Physical examination, self-reported medical history
9. Recent history of significant violence (past 2 years) SCID, Psychiatric Interview
10. Abnormal pseudocholinesterase level Blood testing
11. First degree relative with a psychotic disorder (bipolar disorder, schizophrenia, schizoaffective disorder, or psychosis NOS) SCID, Psychiatric Interview
12. BMI > 35, or a history of documented obstructive sleep apnea Physical examination, self-reported medical history
13. On psychotropic or other medications whose effect could be disrupted by participation in the study Psychiatric interview, self-reported medical history
14. Patients who cannot comply with study procedures during the initial hospitalization phase Study Performance

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: elias dakwar, Principal Investigator — NYSPI
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open-label
Started | 4
Completed | 3
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open-label
Number analyzed (Participants) | 4
Age, Continuous [Mean (Full Range); unit: years] | 50.5 [48 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Use
Description: Participants were provided choices to use up to 5 hits of cocaine on up to 2 occasions (cocaine versus money). Participants who chose cocaine (1 or more hits) during the first choice opportunity are administered a 52 minute infusion of 0.71 mg/kg ketamine the following day. Another choice opportunity occurs 24 hours later. The primary outcome is the choice participants made during these occasions
Time Frame: 5 weeks
Population: medically healthy, treatment-seeking cocaine dependent individuals without a history of abuse of or adverse reaction to ketamine or benzodiazepines.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label
Number analyzed (Participants) | 4
Participants
  first choice opportunity: able to abstain | 3
  first choice opportunity: continue to use | 1
  second choice opportunity: number analyzed (Participants) | 1
  second choice opportunity: able to abstain | 1
  second choice opportunity: continue to use | 0

ADVERSE EVENTS:
Arm/Group | Open-label
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes